CLINICAL TRIAL: NCT05226065
Title: The Relationship Between Intake of Macro and Micronutrients With Clinical Outcomes of Head and Neck Cancer Patients at the Radiotherapy Unit of Dr. Cipto Mangunkusumo Hospital
Brief Title: The Relationship Between Intake of Macro and Micronutrients With Clinical Outcomes of Head and Neck Cancer Patients
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr. Yohannessa Wulandari, M.Gizi, Sp GK, Principal Investigator, Indonesia University
Other Study IDs: 20-08-0928
Record Dates: First submitted 2022-01-06; First posted 2022-02-07 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cancer is a disease caused by uncontrolled cells growth, and its incidence is increasing worldwide. One of the most common cancer is head and neck cancer (HNC), which has low survival rate. Malnutrition occurrence in HNC lower immune system and as result, decreased survival rate was found. Risk factors including tumor histopathology, nutritional status, immune system, and environment have various effects on life expectancy.

Head and neck cancer treatments such as radiotherapy, chemotherapy, and surgery are not without complications. Xerostomia, stomatitis, anorexia, nausea and vomiting, dysgeusia, ageusia, also pain are commonly found during the HNC treatment procedure, and takes part in further undernutrition findings in HNC patients.

Adequate nutrition management has favorable impact in managing HNC patients' malnutrition related problems. Not only energy intake, but also macronutrients and micronutrients intake have been proved be beneficial in the outcomes of HNC patients. Branched-chain amino acids (BCAA) and zinc are namely two nutrients that have been hypothesized to be beneficent. Branched-chain amino acids are found to increase muscle mass, amino acid pools, and immune system, which resulted in preventing malnutrition and cachexia, also increasing total lymphocyte count in cancer patients. Zinc plays role in immune system, antioxidant process, and taste bud functions. Zinc supplementation is correlated to give a better outcome in taste perception and stomatitis in HNC patients who undergo radiotherapy.

This study aims to finds the correlation between BCAA intake with muscle mass and lymphocyte count in HNC patients who haven't undergone chemoradiotherapy, zinc correlation with gustatory in HNC patients who haven't undergone chemoradiotherapy, zinc correlation with stomatitis in HNC patients who is having radiotherapy treatment, and energy and protein intake with body weight in HNC patients after underwent radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* head and neck cancer patients who haven't undergone radiotherapy or chemotherapy, during radiotherapy, and after radiotherapy

Exclusion Criteria:

* have contraindications for body composition measuring
* are immunodeficient or have autoimmune disease
* during immunosuppressant drugs treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Head and neck cancer adult patients who haven't undergone radiotherapy or chemotherapy, during radiotherapy, and after radiotherapy whose came to radiotherapy unit in Dr. Cipto Mangunkusumo Hospital, Jakarta during January 2021 to October 2021.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
body weight | after radiotherapy (1 day)
  body weight in kilogram
total lymphocyte count | before radiotherapy (1 day)
  TLC in 1000/mcL
taste bud perception | before radiotherapy (1 day)
  Henkin test
stomatitis | during radiotherapy (1 day)
  stomatitis grade using WHO criteria
muscle mass | before radiotherapy (1 day)
  body composition analyzer, result in kg.

SECONDARY OUTCOMES:
protein intake | during the first meeting (1 day)
  protein intake using food frequency questionnaire and 24-hrs food recall, data calculated using nutrisurvey
energy intake | during the first meeting (1 day)
  energy intake using food frequency questionnaire and 24-hrs food recall, data calculated using nutrisurvey
BCAA intake | during the first meeting (1 day)
  BCAA intake using food frequency questionnaire and 24-hrs food recall, data calculated using nutrisurvey
zinc intake | during the first meeting (1 day)
  zinc intake using food frequency questionnaire and 24-hrs food recall, data calculated using nutrisurvey
hair zinc level | during the first meeting if the patients undergo radiotherapy (1 day)
  zinc level in hair

CONTACTS AND LOCATIONS:
Overall Officials: Yohannessa Wulandari, MD, Principal Investigator — Indonesia University
Locations (1):
- Dr. Cipto Mangunkusumo Hospital, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

REFERENCES:
- [Derived] Kristian YY, Cahyanur R, Wulandari Y, Sinaga W, Lukito W, Prasetyawaty F, Lestari W. Correlation between branched-chain amino acids intake and total lymphocyte count in head and neck cancer patients: a cross-sectional study. BMC Nutr. 2023 Jul 14;9(1):86. doi: 10.1186/s40795-023-00746-5. PMID 37452428